CLINICAL TRIAL: NCT00381160
Title: Reducing Sugar-Sweetened Beverage Consumption in Overweight Adolescents
Acronym: BASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK73025A; R01DK073025 (NIH)
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Overweight; Obesity
Keywords: weight loss; obesity; sugar-sweetened beverages; diet; adolescence
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

ARMS (2):
- 1 (Experimental): Provision of non-caloric beverages to home
  Interventions: Behavioral: Reduction of sugar-sweetened beverage consumption
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: Reduction of sugar-sweetened beverage consumption — Multi-component intervention aimed at reducing sugar-sweetened beverage consumption. Components include delivery of non-caloric beverages to home in combination with behavioral modification (telephone counseling with parent; check in visit with participant).
  Arms: 1

SUMMARY:
The primary aim of this study is to examine the effect of a multi-component intervention, designed to reduce consumption of sugar-sweetened beverages, on weight gain, total energy intake, and diet quality in adolescents. The secondary aim is to evaluate whether outcomes of the intervention differ between adolescents for whom 100% fruit juice vs. other products (i.e., soda, fruit punch, lemonade, iced tea, coffee drinks, energy drinks, sports drinks) constitutes the primary source of sugar from beverages.

DETAILED DESCRIPTION:
We are partnering with community organizations (including high schools) in the greater Boston area and a major regional supermarket. Participants will be 240 high school students who drink at least 1 serving of sugar-sweetened beverage (including 100% fruit juices) per day and who have a BMI ≥ 85th percentile. They will be randomly assigned to an intervention or control group. The intervention, of 1-year duration, will target the home/family environment in combination with a behavioral intervention provided during brief check-in visits. The environment will be changed by delivering non-caloric beverages to the homes of adolescents who regularly consume sugar-sweetened beverages. Parents will be counseled by telephone to serve as role models in consuming non-caloric beverages. The behavioral intervention for the adolescents will include didactic and experiential components during the check-in visits. Study outcomes will be assessed at baseline, 1 year (end of intervention period), and 2 years (end of follow-up period).

Additional relevant material based on the original proposal (NIH grant application) is provided below:

Each outcome will be compared between groups using a general linear model, adjusted for baseline covariates that could affect body weight: sex, race, ethnicity (Hispanic vs non-Hispanic), household income, parents' education, BMI, beverage consumption (sugar-sweetened, artificially sweetened, unsweetened), energy intake (total, sugar-sweetened beverages, fruit juice), physical activity level, and daily television viewing. Each covariate will be tested for confounding, mediation, and interaction effects on the primary outcome. Stratum-specific estimates of the group difference will be constructed for any covariates showing significant interaction.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in grade 9 or 10
* BMI ≥ 85th percentile for age and gender
* Residing in predominately one household, with access to a working telephone
* Consumption of 12 fluid ounces sugar-sweetened beverages (including 100% fruit juices) per day

Exclusion Criteria:

* Sibling participating in the study
* Intention to change location of residence during the 2 years post-randomization
* Plans to be away from home for 5 weeks or longer during the study period
* Physician diagnosis of a major medical illness or eating disorder
* Chronic use of any medication that may affect body weight or composition
* Current smoking
* Physical, mental, or cognitive handicaps that prevent participation

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2006-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | Change through 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cara B Ebbeing, PhD, Study Director — Boston Children's Hospital; David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ebbeling CB, Feldman HA, Osganian SK, Chomitz VR, Ellenbogen SJ, Ludwig DS. Effects of decreasing sugar-sweetened beverage consumption on body weight in adolescents: a randomized, controlled pilot study. Pediatrics. 2006 Mar;117(3):673-80. doi: 10.1542/peds.2005-0983. PMID 16510646
- [Derived] Ebbeling CB, Feldman HA, Chomitz VR, Antonelli TA, Gortmaker SL, Osganian SK, Ludwig DS. A randomized trial of sugar-sweetened beverages and adolescent body weight. N Engl J Med. 2012 Oct 11;367(15):1407-16. doi: 10.1056/NEJMoa1203388. Epub 2012 Sep 21. PMID 22998339